CLINICAL TRIAL: NCT07196202
Title: Effect of Laid Back Breastfeeding Position on Breastfeeding Experience Among Multiparous Women
Brief Title: Laid Back Breastfeeding Position on Breastfeeding Experience
Acronym: LBB/PBE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Nadia Youssef Ahmed AbdElla, Assistant Professor, Mansoura University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 0669
Record Dates: First submitted 2025-09-19; First posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Maternal Breastfeeding Experience; Maternal Breastfeeding Comfort
Keywords: laid back position; breastfeeding experience; breastfeeding comfort

STUDY DESIGN:
Intervention Model Description: One group of mothers (the intervention group) will be trained on the laid-back position. The other group (the control group) will receive standard care. The outcomes for these two distinct groups were then compared. The groups will treated independently and in parallel.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laid-Back Positioning Group (Active Comparator): Multiparous women who receive structured training and support on the laid-back breastfeeding position during the last trimester of pregnancy so, they can apply it after giving birth
  Interventions: Other: Laid-Back position training
- Standard Care Group (Placebo Comparator): Multiparous women who receive the standard postpartum breastfeeding care and support offered by the hospital after giving birth
  Interventions: Other: Standard Postpartum Care

INTERVENTIONS:
Other: Laid-Back position training — This intervention is a structured training session for pregnant woman on the use of the laid-back breastfeeding position after birth. The training is designed to be delivered in a single, standardized session by the researcher during the last trimester of pregnancy to be applied within the first 24 hours post-cesarean delivery.
  Arms: Laid-Back Positioning Group
Other: Standard Postpartum Care — Postpartum mothers who receive structured training and support on the laid-back breastfeeding position
  Arms: Standard Care Group

SUMMARY:
The goal of this clinical trial is to evaluate the effect of laid back breast feeding position on breastfeeding experience among multiparous women. The main questions it aims to answer are;

* Do postpartum women who feed their babies in a laid-back position report a better breastfeeding experience than those who use the cradle position?
* Do postpartum women who feed their babies in a laid-back position report greater breastfeeding comfort than those who use the cradle position? Researchers will compare breastfeeding in laid-back position to cradle position to see if postpartum women who feed their babies in a laid-back position have better breastfeeding experience and comfort

Participants will:

* Have educational sessions on breastfeeding in laid-back position during antenatal visit of the 3rd trimester
* Will be followed by the researcher for any clarifications about the educational content of session
* Will be asked to apply laid-back position after giving birth, so, the researcher evaluate its effect on breastfeeding experience and comfort.

DETAILED DESCRIPTION:
Cesarean sections are major surgeries that can cause pain and complications, making early breastfeeding initiation less likely compared to vaginal birth. This is problematic because early breastfeeding has significant health benefits for both mother and infant. Breastfeeding outcomes after C-sections are often worse, including delays, more difficulties, and shorter duration.

A common cause of these problems is inadequate breastfeeding technique. The laid-back breastfeeding position is a simple method that relies on the mother's intuition and the baby's natural reflexes, requiring little professional guidance.

This study used a quasi-experimental research design. It will conducted at the antenatal outpatient clinic and inpatient wards of Mansoura University Hospital. The study involved a total of 168 participants. Pregnant mothers in intervention group will be trained to breastfeed their infants using the laid-back position.

ELIGIBILITY:
Inclusion Criteria:

* Multiparous women aged 20 -35 years.
* Multiparous women At the 34 to 36 weeks of gestational age
* Multiparous women with normal course of pregnancy with single-tone fetus
* Multiparous women planning to deliver at Mansoura University Hospital
* Multiparous women who will perform elective caesarian section
* Multiparous women planning to breast feed their babies
* Multiparous women who have no information about laid breastfeeding position
* Multiparous women who will deliver neonate with normal ABGAR score
* Multiparous women who will deliver neonate weight 2.5: 3.5 kg.

Exclusion Criteria:

* Mothers who had inverted or flat nipple.
* Mothers who have postpartum complications
* Mothers who delivered babies with cleft lip, cleft palate, preterm, neurological deficit, asphyxia or any abnormal condition will be excluded from the study.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 168 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Breastfeeding Experience Scale (BES) | 1st time for assessment will be within 24 to 48 hrs after giving birth. 2nd time for assessment will be one week after birth.
  BES consists of 30 items (18- items to assess presence or absence and severity of common breastfeeding difficulties in the early postpartum period and 12 items to assess breastfeeding continuation and the reasons for weaning). In the current study, the researcher used the 18 item part of BES because it suites the aim of the study. The 18-item part are divided into five categories including 3items for breast concern, 5 items for mechanics of breast concern, 5 items for process concern, 3 items for insufficient milk production and 2 items for social concern.
  Scoring system The score system for breastfeeding difficulties using three point Likert scale ranged from "never" (1), "sometimes" (2) and "always" (3). The total scores were ranged from 18 to 54. the level of difficulties were categorized as the following: low severity (< 60%) were ranged from 0 > 32point, average severity (60 % to < 80%) were ranged from 32 > 43 point and high severity (≥80 %) were ranged from 43≥ 54 point.

SECONDARY OUTCOMES:
Maternal comfort during breastfeeding (MCRS) | One week after delivery
  MCRS consists of 9 items describes the maternal feelings during breastfeeding including maternal relaxation during feeding, degree of maternal confidence to hold her baby in laid back position during feeding....ect.
  Scoring system for MCRS The total scores Maternal comfort ranged from 9 to 36 then the level of comfort categorized as; low < 60% (9 - 21); moderate 60% to <75% (22 - 27) & high ≥ 75% (28 - 36).

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Y AbdElla, Asistatnt Professor, Principal Investigator — Faculty of Nursing- Mansoura University- Egypt
Locations (2):
- Egypt (2):
  - Mansoura University Hospitals, Al Mansurah, Dakahlia Governorate
  - New Obstetric and Gynecological Center, Al Mansurah, Dakahlia Governorate

IPD SHARING:
Plan to Share IPD: No
The reason for not sharing data is to comply with and protect the confidentiality of participants, which is a primary ethical requirement in research.